CLINICAL TRIAL: NCT02841332
Title: Multimodal Imaging Analysis of Tissue Changes Occurring During Treatment With Antiangiogenic (Bevacizumab) in Patients With Recurrent Glioblastoma
Brief Title: Multimodal Imaging Analysis During Treatment With Bevacizumab in Patients With Recurrent Glioblastoma
Acronym: IMAGLIO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12 050 03
Record Dates: First submitted 2014-11-03; First posted 2016-07-22 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Glioblastoma
Keywords: Recurrent Glioblastoma; Positron emission tomography; Fluoro misonidazole; MRI multimodal
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with glioblastoma (Experimental): Patient with histologically proved glioblastoma diagnostic will receive the following interventions :
  * Cerebral magnetic resonance imagery
  * Tomography emission positron with F-MISO
  * Bevacizumab administration
  * Clinical examination
  Interventions: Drug: F-MISO; Other: Cerebral magnetic resonance imagery; Drug: Bevacizumab; Other: Clinical examination

INTERVENTIONS:
Drug: F-MISO — The fluoro-misonidazole is a positron emission tomography tracer (labeled with Fluorine-18)-specific hypoxia. This compound penetrates into cells where it is reduced by a nitroreductase enzyme. It is rapidly regenerated by reoxidation when the cell is properly oxygenated. This metabolite can accumulate in viable hypoxic cells (necrotic cells that can provide initial reduction reaction of F-MISO).
  Moreover, the fixing of this tracer appears to be independent of blood flow. The advantage of this technique is to provide a direct image of hypoxic cells by directly targeting under stress hypoxic.
  Other Names: fluoro-misonidazole
Other: Cerebral magnetic resonance imagery — During the pre-therapeutic imagery session :
  * Morphological magnetic resonance imagery ( axial T1 sequence axial T1 post contrast , Flair Axial )
  * magnetic resonance imagery spectroscopy sequence
  * Perfusion magnetic resonance imagery sequence
  * Diffusion magnetic resonance imagery sequence
  Other Names: Cerebral MRI
Drug: Bevacizumab — Administration of bevacizumab during 7 cycles of treatment (J1, J15, J30, J45, J60, J120 and J180)
  Other Names: Avastin
Other: Clinical examination — During the examination, the following parameters will be checked :
  * Neurological examination
  * Corticotherapy prescribed
  * General status of patient (world health organization score)
  * Weight and height
  * Control of arterial pressure
  * Chirurgical and medical history
  * Concomitant treatment

SUMMARY:
The purpose of this study is to estimate the capacity of the multimodal imaging parameters measured at 15 days and 2 months of initiation of treatment with bevacizumab, to measure changes in clinical status (sensitivity to measure changes) in patients treated for recurrent glioblastoma.

DETAILED DESCRIPTION:
Glioblastomas are tumors with poor prognosis. The treatment of recurrent glioblastoma after a standard first-line treatment is not clearly codified, however, many results in the literature show the benefit of bevacizumab (anti- angiogenic therapy) and it is often proposed in this indication . Tissue action, response mechanisms and therapeutic escape remain is poorly understood.

The investigators hypothesize that these response mechanisms are controlled by changes in some parameters in the tumor tissue, such as hypoxia, neoangiogenesis, cell density and that multimodal imaging can help us to better understand these mechanisms.

To identify which parameters of imaging would best measure response mechanisms, the investigators want to evaluate in the first study and for this particular indication , a property of the measure called by the Anglo -Saxon ' sensitivity to change " that is to say, its sensitivity or ability to measure changes. This is an additional property to the reproducibility of the measurement.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization performance index lower or equal to 3
* Estimated life expectancy greater than 3 months
* patient in whom the diagnosis of glioblastoma was histologically proven
* Patient with tumor progression of morphological magnetic resonance imagery evidenced by Pluri Disciplinary Meeting. This increase must meet the detailed criteria Response Assessment Neuro Oncology Working group : except in the case of a new lesion appearing outside of the field of radiotherapy, tumor progression can not therefore be defined on an magnetic resonance imagery performed in a period shorter than 12 weeks after the last day of radiotherapy (see criteria Response Assessment Neuro Oncology Working Group detailed chapter 2-1 B)
* Patient with unilateral tensor above injury at baseline (in order to have in each case a tumor region of interest area and an area equivalent region of interest contralateral healthy tissue) .
* Patient with measurable lesion at baseline, according to the criteria defined by the working group Respons Assessment Neuro Oncology. The lesion with contrast is measured two-dimensionally on T1 gadolinium in axial section. The two perpendicular diameters of red lead should be 10 mm and that at least two axial sections.
* Patient with progression after radiotherapy and have received at least one chemotherapy regimen (temodal)
* A patient in whom treatment with bevacizumab monotherapy

Exclusion Criteria:

* Pregnancy
* Exclusion criteria related to cons to the realization of positron emission tomography or magnetic resonance imagery : Weight greater than 120 kg, Foreign body incompatible with magnetic resonance imagery (eg metallic intraocular foreign body), Medical equipment installed incompatible with magnetic resonance imagery (eg pacemaker)
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Detection capacity of patient clinical status in imagery with F-MISO as assessed by tomography with emission of positron | At day 15 after the 1st perfusion of bevacizumab
  Specific imagery parameters used are :
  Standard Uptake Value max, mean Standard Uptake Value, global or tumoral volume reported
Detection capacity of patient clinical status in imagery with F-MISO as assessed by Perfusion magnetic resonance imagery | At day 15 after the 1st perfusion of bevacizumab
  Specific imagery parameters used are :
  Cerebral blood volume and relative cerebral blood volume, absolute neo angiogenesis and reported to tumoral volume
Detection capacity of patient clinical status in imagery with F-MISO as assessed by Diffusion magnetic resonance imagery | At day 15 after the 1st perfusion of bevacizumab
  Specific imagery parameters used are :
  Apparent diffusion Coefficient and Apparent diffusion relative Coefficient , absolute elevated cellular density volume and reported to tumoral volume
Detection capacity of patient clinical status in imagery with F-MISO as assessed by Spectroscopy magnetic resonance imagery | At day 15 after the 1st perfusion of bevacizumab
  Specific imagery parameters used are :
  choline pike, NAA pike, mean and maximal creatinine pike, mean and maximal ratio choline/NAA, mean and maximal ratio choline/creatinine
Detection capacity of patient clinical status in imagery with F-MISO as assessed by tomography with emission of positron | At day 60 after the 4th perfusion of bevacizumab
  Specific imagery parameters used are :
  Standard Uptake Value max, mean Standard Uptake Value, global or tumoral volume reported
Detection capacity of patient clinical status in imagery with F-MISO as assessed by Perfusion magnetic resonance imagery | At day 60 after the 4th perfusion of bevacizumab
  Specific imagery parameters used are :
  Cerebral blood volume and crelative cerebral blood volume, absolute neo angiogenesis and reported to tumoral volume
Detection capacity of patient clinical status in imagery with F-MISO as assessed by Diffusion magnetic resonance imagery | At day 60 after the 4th perfusion of bevacizumab
  Specific imagery parameters used are :
  Apparent diffusion Coefficient and Apparent diffusion relative Coefficient , absolute elevated cellular density volume and reported to tumoral volume
Detection capacity of patient clinical status in imagery with F-MISO as assessed by Spectroscopy magnetic resonance imagery | At day 60 after the 4th perfusion of bevacizumab
  Specific imagery parameters used are :
  choline pike, NAA pike, mean and maximal creatinine pike, mean and maximal ratio choline/NAA, mean and maximal ratio choline/creatinine

SECONDARY OUTCOMES:
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with relative cerebral blood volume in Perfusion magnetic resonance imagery | at day 15 after the 1st perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with relative cerebral blood volume in Perfusion magnetic resonance imagery | at day 60 after the 4th perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with apparent diffusion coefficient on diffusion magnetic resonance imagery | at day 15 after the 1st perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with apparent diffusion coefficient on diffusion magnetic resonance imagery | at day 60 after the 4th perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with rate of choline on spectroscopy magnetic resonance imagery | at day 15 after the 1st perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with rate of choline on spectroscopy magnetic resonance imagery | at day 60 after the 4th perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with rate of N-acetyl aspartate on spectroscopy magnetic resonance imagery | at day 15 after the 1st perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with rate of N-acetyl aspartate on spectroscopy magnetic resonance imagery | at day 60 after the 4th perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with rate of rate of creatinine on spectroscopy magnetic resonance imagery | at day 15 after the 1st perfusion of bevacizumab
Estimation of predictive parameters of progression free survival with a sensibility of change of at least 75% as assessed with rate of rate of creatinine on spectroscopy magnetic resonance imagery | at day 60 after the 4th perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by relative cerebral blood volume in Perfusion magnetic resonance imagery | At day 15 after the first perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by relative cerebral blood volume in Perfusion magnetic resonance imagery | At day 60 after the 4th perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by apparent diffusion coefficient on diffusion magnetic resonance imagery, | At day 15 after the 1st perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by apparent diffusion coefficient on diffusion magnetic resonance imagery, | At day 60 after the 4th perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by rate of choline on spectroscopy magnetic resonance imagery | At day 15 after the 1st perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by rate of choline on spectroscopy magnetic resonance imagery | At day 60 after the 4th perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by N-acetyl aspartate on spectroscopy magnetic resonance imagery | At day 15 after the 1st perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by N-acetyl aspartate on spectroscopy magnetic resonance imagery | At day 60 after the 4th perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed byrate of creatinine on spectroscopy magnetic resonance imagery | At day 15 after the 1st perfusion of bevacizumab
Estimation of imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% as assessed by rate of creatinine on spectroscopy magnetic resonance imagery | At day 60 after the 4th perfusion of bevacizumab
Variation in imagery predictive parameters for progression free survival with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by relative cerebral blood volume in Perfusion magnetic resonance imagery | At day 15 and day 60
Variation in imagery predictive parameters for progression free survival with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by apparent diffusion coefficient on diffusion magnetic resonance imagery | At day 15 and day 60
Variation in imagery predictive parameters for progression free survival with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by rate of choline on spectroscopy magnetic resonance imagery | At day 15 and day 60
Variation in imagery predictive parameters for progression free survival with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by N-acetyl aspartate on spectroscopy magnetic resonance imagery | At day 15 and day 60
Variation in imagery predictive parameters for progression free survival with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by rate of creatinine on spectroscopy magnetic resonance imagery | At day 15 and day 60
Variation in imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by relative cerebral blood volume in Perfusion magnetic resonance imagery | At day 15 and day 60
Variation in imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by apparent diffusion coefficient on diffusion magnetic resonance imagery | At day 15 and day 60
Variation in imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by rate of choline on spectroscopy magnetic resonance imagery | At day 15 and day 60
Variation in imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by rate of N-acetyl aspartate on spectroscopy magnetic resonance imagery | At day 15 and day 60
Variation in imagery prognostic parameters for global survival at 6 months with a sensibility of change of at least 75% between cycle 1 and cycle 4 of treatment as assessed by rate of creatinine on spectroscopy magnetic resonance imagery | At day 15 and day 60

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Benouaich-Amiel, MD, Principal Investigator — U H Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No